CLINICAL TRIAL: NCT04122690
Title: Partnered Dance Aerobic Exercise as a Neuroprotective, Motor and Cognitive Intervention in Parkinson's Disease
Acronym: PDAE in PD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: F2967-R; IRB112770 (Other Grant/Funding Number: United States Department of Affairs)
Record Dates: First submitted 2019-10-09; First posted 2019-10-10 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Parkinson's Disease; Exercise Therapy; Cognition
Keywords: motor control; Parkinson disease; exercise; neural imaging; dance; spatial cognition; executive function; substantia nigra; neurodegeneration; rehabilitation
MeSH Terms: conditions — Parkinson Disease; Motor Activity; Nerve Degeneration

STUDY DESIGN:
Intervention Model Description: PDAE compared with WAE
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Partnered Dance Aerobic Exercise (Experimental): Partnered Dance-Aerobic Exercise (PDAE) is an adapted form of Argentine tango, aka Adapted tango. Participants with PD will dance the follower role only and will dance with new partners (individuals without PD) every 15-20 minutes, a widely practiced method considered by the dance teaching community to enhance learning. Participants will engage in partnering exercises on how to interpret motor goals through touch, exercises to develop understanding of temporal relationship of movement to music, novel step introduction, connecting previously learned and novel step elements. Frequent repetition and musical stereotypes may foster implicit learning or muscle memory (i.e., motor learning, or procedural memory that involves consolidating a specific motor task into memory through repetition). Participants will not be required to memorize specific step patterns but will learn new steps in each class
  Interventions: Behavioral: PDAE
- Walking Aerobic Exercise (Active Comparator): Walking Aerobic Exercise (WAE) Participants in WAE will receive equivalent dose, volume, frequency, intensity and duration of exercise to the PDAE group. The investigators will receive equal contact and monitoring from study staff. WAE participants will report to the same facility and interact with the same interventionist and assistants. The investigators will participate in sessions focused on at least 60 minutes of walking with breaks ad libitum, and 1/2 hour balance and stretching. The investigators have a designated, safe and non-cluttered area for walking. WAE will also take place in groups, with research volunteers and assistants to ensure that PDAE and WAE participants both receive a socially engaging intervention.
  Interventions: Behavioral: WAE

INTERVENTIONS:
Behavioral: PDAE — Participants with PD will dance the follower role only and will dance with new partners (individuals without PD) every 15-20 minutes, a widely practiced method considered by the dance teaching community to enhance learning. Participants will engage in partnering exercises on how to interpret motor goals through touch, exercises to develop understanding of temporal relationship of movement to music, novel step introduction, connecting previously learned and novel step elements. Frequent repetition and musical stereotypes may foster implicit learning or muscle memory (i.e., motor learning, or procedural memory that involves consolidating a specific motor task into memory through repetition). Participants will not be required to memorize specific step patterns but will learn new steps in each class
  Arms: Partnered Dance Aerobic Exercise
Behavioral: WAE — The participants will receive equal contact and monitoring from study staff. WAE participants will report to the same facility and interact with the same interventionist and assistants. The participants will participate in sessions focused on at least 60 minutes of walking with breaks ad libitum, and 1/2 hour balance and stretching. The investigators have a designated, safe and non-cluttered area for walking. WAE will also take place in groups, with research volunteers and assistants to ensure that PDAE and WAE participants both receive a socially engaging intervention
  Arms: Walking Aerobic Exercise

SUMMARY:
Parkinson's disease (PD) is a difficult to treat condition that impairs mobility and thinking. It is not fully treated by drugs and surgery. Two priority issues for most people with PD are "OFF-time" and Cognitive impairment. Even under best medical management, 74% of people with PD experience "OFF-time," which is when medications are just not working right. OFF-time severely impacts both quality of life and thinking. Cognitive problems are found even in newly diagnosed people with PD and are very difficult to treat. However, the investigators' research has shown that partnered dance-aerobic exercise (PDAE) reduces OFF-time on the official test for OFF-time of the Movement Disorders Society, the Movement Disorders Society Unified Parkinson Disease Rating Scale-IV, (MDS-UPDRS-IV). PDAE improves other symptoms too. Benefits of the therapy have lasted for at least one-month after PDAE sessions stopped. PDAE provides aerobic exercise during an improvisational, cognitively-engaging physical activity. Cognitive engagement is a critical component of PDAE. Previous research showed PDAE improved spatial cognition, the ability to navigate, to mentally picture shapes and paths in the mind and to know the relationships between objects, people and places. Also, the investigators showed with imaging of the brain using a magnet in a scanner that twice weekly PDAE training increases activity in brain regions used in thinking and decision making. The investigators know that exercise benefits mobility and cognitive problems. The investigators even think exercise might protect brain cells in people with PD. But no one has really been able to show with biomarkers that exercise is protective of brain cells in humans.

DETAILED DESCRIPTION:
The investigators will conduct a study in Veterans and non-Veterans with diagnosed PD to compare PDAE versus walking for OFF-time, cognition, and brain cell protection. The investigators will use a method like a coin flip to decide if the participants will be doing PDAE or walking. Importantly, the investigators will see if brain cells are protected using a brain scan that looks at the areas affected by PD to determine the relative amounts of different hormones in the brain that are related to having Parkinson's. The investigators will use these measurements of these hormones to chart the course of brain cell breakdown in patients with PD who have done walking or PDAE for 16 months. The investigators think that that PDAE will be better at lessening OFF-time and making cognition better than walking. The investigators think this because participants have to really use the mind during PDAE because the participants have so much to think about in terms of the steps and patterns. The investigators will assign 102 Veterans with mild-moderate PD to either 16 months of PDAE or walking. The investigators will use a coin toss or other similar method to determine who goes in what group. The investigators need participants to be in the classes for 16-months because it takes that long for us to see if anything changed in the brain with those hormones. Participants will do twice weekly classes for the first 3 months and then will switch down to taking lessons just 1 time per week for 13 months. The investigators will schedule appointments for participants to be seen by the research team before Veterans begin lessons, at 3 months (after the twice weekly schedule) and at 16 months after all the lessons are completed. The appointments will consist of asking the Veterans about their OFF-time having them take a few memory and thinking tests. The investigators will also ask them to lie in a scanner for about an hour. The participants can rest in the scanner for about a 1/2 hour and also do a thinking task. The investigators will be able to answer the questions, "Is PDAE better than walking at lessening OFF-time and spatial cognition and slowing down brain cell death? This study is using cutting edge imaging techniques for the first time to see if dance or walking are helpful for slowing brain cell death. This project combines patient-centered, clinical science and mechanistic aims to improve health care.

ELIGIBILITY:
Inclusion Criteria:

* Age: older than 40 years (40 is upper limit for young onset PD)
* Montreal Cognitive Assessment (MoCA) score >17
* Able to walk with or without an assistive device at least 10 feet
* Best corrected/aided acuity better than 20/70 in the better eye
* Willingness to be randomized to either group
* H&Y stages I-III
* Report OFF times (reporting >0 on item 4.3 of the UPDRS-IV)
* Show clear symptomatic benefit from antiparkinsonian medications

  * e.g., alleviated rigidity, bradykinesia, and tremor
* Fluent in English to comprehend and participate

Exclusion Criteria:

* Untreated Major Depression and major psychiatric illness
* History of stroke, or traumatic brain injury
* Pure-tone threshold average sensitivity at 0.5, 1.0, and 2.0 kHz exceeds 40 dB
* Previous participation in PDAE or WAE classes.
* Alcohol abuse and/or use of antipsychotics
* Lives outside of the study site or is planning to move out of the area in next year or leave the area for >1 month during the next year
* Taking moderate to high doses of beta-blockers with a resting heart rate below 60 beats/min since exercise intensity is measured through target heart rate.
* Severe cardiac disease, including:

  * New York Heart Association (NYHA) Class III or IV congestive heart failure
  * clinically significant aortic stenosis
  * history of cardiac arrest, use of a cardiac defibrillator
  * uncontrolled angina

    * as discussed we are not planning to perform routine exercise tolerance tests prior to enrollment
* Other significant co-morbid disease that would impair ability to participate in the exercise-based intervention

  * e.g. renal failure on hemodialysis, excessive alcohol use (>14 drinks per wk)
* Any contraindications to MRI eg claustrophobia, etc

Ages: 40 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2021-01-25 (Actual); Primary Completion 2026-12-15 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
Movement disorders Society Unified Parkinson's Disease Rating Scale Part IV total score | 16 months
  The primary outcome, the MDS-UPDRS-IV score measures medication related motor fluctuations, including dyskinesias, OFF-time, functional impact and complexity of fluctuations, and dystonia. The investigators will administer a monthly OFF-state diary for corroboration of these scores.
Corsi Blocks product score | 16 months
  The product score is the product of the span and number of correct trials achieved by the participant. The Corsi Blocks is a test of spatial cognition, specifically visuospatial working memory.
rate of change in iron accumulation in the substantia nigra pars compacta | 16 months
  The investigators will measure R2* in the NM-MRI defined SNc using a published image processing and analysis method. This method leverages a standard space SNc atlas developed using control population NM-MRI data, enabling R2* measurement in SNc with no operator-dependent segmentation steps

SECONDARY OUTCOMES:
6 minute walk test (number of meters walked in 6 minutes) | 16 months
  The six minute walk test is a validated test of endurance in older adults and in those with Parkinson disease. Participants are asked to walk as far as they can in 6 minutes, while being monitored and able to carry on a conversation. The distance is measured in meters.
cardiovascular output: V02 maximum | 16 months
  This sub-maximal test can estimate the participant's VO2max and initial fitness level. This test uses a method in which heart rate (HR) workload values are obtained at 2-4 points and extrapolated to predict workload at the estimated maximum HR (e.g. 220-age). VO2max is then calculated from the predicted maximum workload.
neural measure of spatial cognition (BOLD signal) | 16 months
  At each study visit T1 MPRAGE, and T2* weighted blood oxygen level dependent (BOLD) fMRI data will be acquired at the Emory CSI, using a Siemens Prisma-Fit 3T MRI scanner with a 64 channel receive-only head coil in a protocol with total scan time one hour. BOLD signal will be measured in response to the functional task, the Block span task.
rate of change in loss of neuromelanin in substantia nigra pars compacta | 16 months
  At each study visit NM-MRI, R2*, T1 MPRAGE, and T2* weighted blood oxygen level dependent (BOLD) fMRI data will be acquired. The investigators will carry out image processing to determine SNc volume using an automated approach previously shown to have high scan-rescan reproducibility.
Executive function: Tower Of London achievement score | 16 months
  The Delis Kaplan tower of London test is a validated measure of executive function in PD.
Benton's judgment of line orientation task | 16 months
  Judgment of Line Orientation is a standardized test of visuospatial skills commonly associated with functioning of the parietal lobe in the right hemisphere. The test measures a person's ability to match the angle and orientation of lines in space. Subjects are asked to match two angled lines to a set of 11 lines that are arranged in a semicircle and separated 18 degrees from each other.
gait- forward, fast as possible, backward speeds | 16 months
  Objective, spatiotemporal parameters including velocity, stride length, stance percent, velocity variability and other variables of preferred, backward and fast-as-possible walking will be assessed.
attention: Trails Making Test A | 16 months
  Trails making test A is a validated measure of attention and visuospatial processing in people with PD. The time to complete is considered.
spatial imagery: Brooks spatial memory task percent correct | 16 months
  Brooks spatial memory involves reporting back a specified path of numbers that patients are asked to visualize in a 4 x 4 grid.

OTHER OUTCOMES:
Mini BESTest score | 16 months
  The Mini BESTest is a 14-item test scored on a 3-level ordinal scale. Mini BESTest assesses dynamic balance, a unidimensional construct. It is validated in PD.
Four Square Step Test (time to complete) | 16 months
  The FSST is a valid measure of motor cognitive integration and involves the participant stepping as quickly and safely as they can in four quadrants created by four canes arranged in a cross, in a clockwise order and then switching to counterclockwise order.
Dynamic Gait index | 16 months
  The DGI is a clinical tool to assess gait, balance and fall risk. It evaluates not only usual steady-state walking, but also walking during more challenging tasks.
Single/Dual Timed up and go (time to complete and dual task costs) | 16 months
  Timed Up & Go Test (TUG) is a test of balance that is commonly used to examine functional mobility. The single condition requires participants to get up from a chair walk three meters, turn around and return to the chair as quickly and as safely as they can. The dual versions involve cognitive tasks (counting backward by 3s from given number) and manual, holding a full cup of water, while performing single tug.
Parkinson Disease Questionnaire -39 | 16 months
  The PDQ-39 is a 39-item self-report questionnaire, which assesses Parkinson's disease-specific health related quality over the last month Assesses how often patients experience difficulties across the 8 quality of life dimensions
composite physical function index | 16 months
  This validate scale assesses the ability of people with impairments to complete various tasks of daily living ranging from holding a bag of groceries to walking a couple of blocks to being able to take a bath unassisted.
Movement disorders Society Unified Parkinson's disease rating scale parts I-III | 16 months
  Part I assesses non motor aspects of experiences of daily living for people with PD. Part II assesses motor aspects of experiences of daily living for people with PD. Part III is a rated scale of motor function. The MDS UPDRS is validated and reliable and widely used globally.
Beck depression inventory score | 16 months
  This widely used test of depression is validated in PD.
Freezing of Gait questionnaire total score | 16 months
  The Freezing of Gait Questionnaire (FOG-Q) reliably detects FOG in patients with Parkinson's disease (PD).
Physical Scale for the Elderly score (PASE) | 16 months
  PASE comprises measures of self-reported occupational, household, and leisure activities during a one-week period. Designed for use in epidemiologic studies and exercise interventions, the instrument can be administered by telephone, mail, or in person in 5 to 15 minutes.
Short Form 12 | 16 months
  A generic, multipurpose short-form survey with 12 questions selected from the SF-36 Health Survey which, when combined, scored and weighted, results in two scales of mental and physical functioning and overall health-related quality of life. Subscales of interest include the Mental composite and physical composite scores among others.
Satisfaction with Training period questionnaire | 3 months
  Participants will complete the Exit Questionnaire which asks their level of agreement on a Likert scale (1-5) with 1 indicating the most agreement about whether they think they improved in various aspects of wellbeing.
Satisfaction with Maintenance period questionnaire | 16 months
  Participants will complete the Exit Questionnaire which asks their level of agreement on a Likert scale (1-5) with 1 indicating the most agreement about whether they think they improved in various aspects of wellbeing.
Satisfaction with Life scale | 16 months
  Valid for PD, this scale allows self report of level of satisfaction with life and life events in people with PD.
Multidimensional Scale of Perceived social support (MSPSS) | 16 months
  The MSPSS aims to determine how social support factors are perceived by individuals, with three subscales to evaluate support by family, friends and significant others.

CONTACTS AND LOCATIONS:
Overall Officials: Madeleine E. Hackney, PhD, Principal Investigator — Atlanta VA Medical and Rehab Center, Decatur, GA
Locations (1):
- Atlanta VA Medical and Rehab Center, Decatur, GA, Decatur, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim H, Rafie F, Nekouei AH, Kazanski ME, Hackney ME. Compliance and Satisfaction for 16 months of Adapted Tango vs. Supervised Walking for People with Parkinson's. NPJ Parkinsons Dis. 2025 Dec 26;12(1):13. doi: 10.1038/s41531-025-01220-8. PMID 41453883
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2024 Apr 8;4(4):CD013856. doi: 10.1002/14651858.CD013856.pub3. PMID 38588457
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 Jan 5;1(1):CD013856. doi: 10.1002/14651858.CD013856.pub2. PMID 36602886

DOCUMENTS (1):
  • Informed Consent Form (2021-12-16): https://cdn.clinicaltrials.gov/large-docs/90/NCT04122690/ICF_000.pdf